CLINICAL TRIAL: NCT03905759
Title: Preoperative Colchicine, Dronedarone Or Amiodarone for Prophylaxis Against Postoperative Atrial Fibrillation in Patients Undergoing On-pump CABG; A Comparative Study
Brief Title: Prophylaxis Against Postoperative Atrial Fibrillation in Patients Undergoing On-pump CABG
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: doaa rashwan (Other)
Responsible Party: Sponsor-Investigator, doaa rashwan, Assistant profesor Doaa Rashwan, Beni-Suef University
Organization: Beni-Suef University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: FMBSURECS/31032019/Mohammed
Record Dates: First submitted 2019-04-01; First posted 2019-04-05 (Actual); Last update posted 2019-04-05 (Actual); Status verified 2019-04

CONDITIONS: Postoperative Atrial Fibrillation
MeSH Terms: interventions — Dronedarone; Amiodarone; Colchicine

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- colchicine (Active Comparator): Colchicine will be used at the dose of 1 mg orally, twice daily, preoperatively (1 days), and of 0.5 mg, twice daily, until hospital discharge
  Interventions: Drug: Colchicine
- Dronedarone (Active Comparator): Dronedarone (200 mg twice daily starting from day before operation till 5 days after)
  Interventions: Drug: Dronedarone
- amiodarone (Active Comparator): amiodarone (200 mg three times per day)21 administered 6 days prior to surgery through 6 days after surgery
  Interventions: Drug: Amiodarone

INTERVENTIONS:
Drug: Dronedarone — Dronedarone (200 mg twice daily starting from day before operation till 5 days after)
  Other Names: amiodarone,colchicine
  Arms: Dronedarone
Drug: Amiodarone — Group A:-amiodarone (200 mg three times per day)21 administered 6 days prior to surgery through 6 days after surgery
  Other Names: colchicine ,dronedarone
  Arms: amiodarone
Drug: Colchicine — Colchicine will be used at the dose of 1 mg orally, twice daily, preoperatively (1 days), and of 0.5 mg, twice daily, until hospital discharge
  Other Names: amiodarone, dorendarone
  Arms: colchicine

SUMMARY:
Atrial fibrillation in the postoperative period of myocardial revascularization surgery (AF-POMR) occurs in 10% to 65% of patients, increasing morbidity and mortality after surgery. is associated with an increase in hospital length of stay, and, thus, in costs,and can cause serious clinical complications, such as hypotension, heart failure, stroke and other thromboembolic disorders.Although not completely understood, the electrophysiological mechanism of AF-POMR is believed to be reentry.

DETAILED DESCRIPTION:
Aim of the study The aim of this work is to study the effect of preoperative Colchicine, Dronedarone or Amiodarone for prophylaxis against postoperative atrial fibrillation in patients undergoing on-pump CABG.

Patients and Methods

Type and site of the study:

This randomized double blinded clinical study will be carried out at Beni-Suef university hospital, after approval by the department of Anesthesiology, Pain management and Surgical ICU, the local ethics and research committee and other involved departments, faculty of medicine, Beni-Suef University.

Study population:

The study population will include inpatients of the cardiothoracic department scheduled for CABG surgery, both sex, selected randomly according to American Society of Anesthesiologists(ASA) grade II and III, between the ages of 40 -60ears.

Exclusion criteria:.

* Liver dysfunction, pregnancy.
* History of allergic reaction to any drug used in this study.
* Emergency procedure
* Preoperative dialysis
* A.F.
* Patients on antiarrhythmic medications

Sample size estimation:

As considered the primary outcome, sample size calculation was done using the comparison of the rate of occurrence of postoperative AF in cases undergoing on-pump CABG pretreated with colchicine, dronedarone or amiodarone. As previously published 19 , the rate of postoperative AF among amiodarone group was 25%, while in colchicine, it was 7% 20. investigators assumed that dronedarone treatment will differ about 20% from amiodarone and selected the least excepted difference to do the calculation. Therefore, the calculation was done based on comparing 2 proportions from independent samples using Chi test, the α-error level was fixed at 0.05 and the power was set at 80%.

Accordingly, the optimum sample size should be 48 cases in each arm. Sample size calculation was done using PS Power and Sample Size Calculations software, version 3.0.11 for MS Windows (William D. Dupont and Walton D. Vanderbilt, USA).

Sampling Technique:

The patients will be randomly divided into three groups, as follows: Group c: Colchicine will be used at the dose of 1 mg orally, twice daily, preoperatively (1 days), and of 0.5 mg, twice daily, until hospital discharge ; Group D: Dronedarone (200 mg twice daily starting from day before operation till 5 days after) ; Group A:-amiodarone (200 mg three times per day)21 administered 6 days prior to surgery through 6 days after surgery Randomization assignment of patients to Groups C, D and A will be performed with a list of random numbers generated by a computer program's random function. The allocation into the groups and the preparation of the study drug will be performed by an individual who as unrelated to the study. Personnel, patients, and the individual participating in the data collection and data analysis will be blinded to the treatment assignments.

Anesthesia Management The patients will be evaluated preoperatively 1 day before surgery. Electrocardiogram (ECG), pulse oximetry, cannulation of the invasive arterial pressure (20 gauge) from the left radial artery, and peripheral venous access (18 gauge) from the right arm will be inserted into the patient, who will be taken to the operating room on the day of the surgery. After induction of anesthesia and intubation, an 8F central venous catheter will be inserted from the right internal jugular vein. Midazolam (0.05 mg/kg), propofol (2 mg/kg), fentanyl (5 mcg/kg), and rocuronium (0.6 mg/kg) will be used for the induction of anesthesia. Anesthesia will be maintained with a mixture of 2% sevoflurane, 60% oxygen, and 40% air.

All patients will be ventilated with positive pressure. Ventilation parameters will be set as a tidal volume of 8ml/kg and a respiratory rate of 10-12/min, which will be assessed by arterial blood gases. All patients will receive 500 ml ringer lactat before the induction of anesthesia. Thereafter, IV ringer lactate solution will be infused to keep the central venous pressure (CVP) at 10-12 mmHg.

Cardiopulmonary Bypass Management Before cannulation for CPB, 3 mg/kg of heparin will be administered for all patients. When the activated coagulation time will be > 400/sec, it will be passed to the pump.

Nonpulsatile CPB flow rates of 2-2.4 L/min/m2 will be applied, and the mean arterial pressure (MAP) will be kept at 50-60 mmHg. Hematocrit concentration will be maintained at 25-28%. Moreover, mild hypothermia (28-30°C) will be reached during CPB. Myocardial protection will be achieved with intermittent antegradecardtemperature of 37°C will be achieved after surgery, and the patient will be removed from CPB. Following this, coagulation will be provided with protamine; once hemodynamic stabilization (MAP 70-90 mmHg) will be achieved, patients will be brought to the intensive care unit.

Data Collection Methods:

The following parameters will be evaluated and recorded by senior anesthesiologist unaware of the study protocol:

* Demographic data (age, sex, and weight)
* Perioperative data (operation time, cross-clamp time, EF ).
* Post bypass and post operative AF
* Hospital stay and death

Statistical analysis Continuous variables will be summarized as mean ± SD and categorical variables Will be expressed as proportion (%). Univariate analyses will be performed by chi-square, student's t-test, Fisher exact test, Mann Whitney test and One-way ANOVA (will be used for comparison between the three groups). SPSS for Windows (version 17; SPSS Inc., Chicago, IL., USA) will be used for statistical analysis. Results will be considered significant if P values are less than 0.05p

ELIGIBILITY:
Inclusion Criteria:

The study population will include inpatients of the cardiothoracic department scheduled for CABG surgery, both sex, selected randomly according to American Society of Anesthesiologists(ASA) grade II and III

Exclusion Criteria:

* - Liver dysfunction, pregnancy.
* History of allergic reaction to any drug used in this study.
* Emergency procedure
* Preoperative dialysis
* A.F.
* Patients on antiarrhythmic medications

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 48 (Estimated)
Dates: Start 2019-04-03 (Actual); Primary Completion 2020-04-10 (Estimated); Study Completion 2020-04-10 (Estimated)

PRIMARY OUTCOMES:
AF | change from baseline rhythm at 6 days
  incidence of AF

CONTACTS AND LOCATIONS:
Overall Officials: belal Y Mohammed, Msc, Principal Investigator — Faculty of Medicine Beni-Suef University
Locations (1):
- Faculty Of Medicine, Beni-Suef University, Banī Suwayf, Egypt

IPD SHARING:
Plan to Share IPD: Yes
the protocol
Supporting Information: Study Protocol
Time Frame: after registration for ever
Access Criteria: on the web page